CLINICAL TRIAL: NCT00164996
Title: Comparison of Ultrathin Versus Conventional Esophagogastroduodenoscopy in Unsedated Patients With or Without Local Pharyngeal Anaesthesia: A Randomized Controlled Trial
Brief Title: Ultrathin Versus Conventional Esophagogastroduodenoscopy in Unsedated Patient With or Without Local Pharyngeal Anaesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE 2004.312
Record Dates: First submitted 2005-09-10; First posted 2005-09-14 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2005-09

CONDITIONS: Dyspepsia
Keywords: upper endoscopy; local pharyngeal anaesthesia; ultrathin endoscope
MeSH Terms: conditions — Dyspepsia

INTERVENTIONS:
Procedure: Local pharyngeal anaesthesia
Device: Ultrathin endoscope

SUMMARY:
The purpose of this study is to investigate whether an ultrathin endoscope will improve a patient's tolerance during the procedure. In addition, this study will look at whether local pharyngeal anaesthesia is necessary during ultrathin endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-70

Exclusion Criteria:

* Previous experience of upper endoscopy
* Allergy to local pharyngeal anaesthesia
* Patient requesting sedation during endoscopy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2004-09; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
patient's tolerance and anxiety in visual analog scale (VAS) score

SECONDARY OUTCOMES:
patient's satisfaction; procedure time; complications

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Lik-Man Mui, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, China